CLINICAL TRIAL: NCT05989633
Title: DERCOS DS DANDRUFF TREATMENT OBSERVATIONAL STUDY 2022
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: Dercos DS in Dandruff
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Dandruff
Keywords: dandruff; treatment satisfaction
MeSH Terms: conditions — Dandruff

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dermocosmetic product: Selenium Disluphide Shampoo (Dercos DS) — to assess the benefit of Dercos DS in subjects with dandruff

SUMMARY:
The aim of this study is to evaluate the satisfaction / tolerance / cosmeticity of Dercos DS

ELIGIBILITY:
Inclusion Criteria:

* Patients with dandruff or seborrheic dermatitis
* All hair types
* All ethnicities (Asian, Caucasian, Afro-American, African, Hispanic)
* Including patients with specific occlusion habits (for instance veil use at least 8 hours per day, hat use)
* Patients willing to provide written informed consent

Exclusion Criteria:

* Under 12 years old
* Pregnancy, breast feeding, childbearing potential without adequate contraception, or irregular menstrual cycles.
* History of allergy, anaphylaxis or hypersensitivity to any of the ingredients of Shampoo any of the ingredients of DERCOS ANTI-DANDRUFF normal to oily hair shampoo
* History of allergic contact dermatitis secondary to shampoo, conditioner, mask, and/or leave-in.
* Has any clinical manifestations in the treatment(s) or other disorders that, in the opinion of the investigator, may affect the evaluations or results of the study products.- Inability to stay the study period (56 days +-5 days) without performing any hair/scalp procedure, including coloring, straightening and cutting.
* Inability to attend all study visits and follow treatment regimen

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with dandruff or seborrheic dermatitis
Sampling Method: Non-Probability Sample
Enrollment: 5131 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Desquamation | Baseline
  Scale (0=absence to 4= very severe)
Desquamation | Day 28
  Scale (0=absence to 4= very severe)
Desquamation | Day 56
  Scale (0=absence to 4= very severe)
Irritation | baseline
  Scale (0=absence to 4= very severe)
Irritation | Day 28
  Scale (0=absence to 4= very severe)
Irritation | Day 56
  Scale (0=absence to 4= very severe)
Erythema | baseline
  Scale (0=absence to 4= very severe)
Erythema | Day 28
  Scale (0=absence to 4= very severe)
Erythema | Day 56
  Scale (0=absence to 4= very severe)
Itching | baseline
  Scale (0=absence to 10= very severe)
Itching | Day 28
  Scale (0=absence to 10= very severe)
Itching | Day 56
  Scale (0=absence to 10= very severe)
Area involved | baseline
  scale from <10% to >90%
Area involved | Day 28
  scale from <10% to >90%
Area involved | Day 56
  scale from <10% to >90%
Tolerance | baseline
  scale from 0= none to 5=very tolerated
Tolerance | Day 28
  scale from 0= none to 5=very tolerated
Improvement | Day 28
  scale from 0= worse to 5=very clearly improved
Improvement | Day 56
  scale from 0= worse to 5=very clearly improved
Impact of dandruff on patient | baseline
  Scale from 0=not bothered at all to 5=very bothered
Impact of dandruff on patient | Day 28
  Scale from 0=not bothered at all to 5=very bothered
Impact of dandruff on patient | Day 56
  Scale from 0=not bothered at all to 5=very bothered
Global evaluation by investigator | Day 28
  Scale from 0=not at all satisfactory at all to 4=very satisfactory
Global evaluation by investigator | Day 56
  Scale from 0=not at all satisfactory at all to 4=very satisfactory
Assessment of hair fiber and quality | Day 56
  scale from 0=worsened to 4=very improved
Product respect/protects hair fiber | Day 56
  scale from 0=no, it is now more damaged/dry than before the treatment to 3=Yes, my hair fiber looks/feels better than before the treatment
Patient product efficacy satisfaction | Day 28
  questionnare with scale ranging from 0=completely disagree to 5=completely agree
Patient product efficacy satisfaction | Day 56
  questionnare with scale ranging from 0=completely disagree to 5=completely agree
Patient product acceptability | Day 28
  scale ranging from 0=not satisfied at all to 10=very satisfied
Patient product acceptability | Day 56
  scale ranging from 0=not satisfied at all to 10=very satisfied
Patient global satisfaction | Day 28
  scale ranging from 0=not satisfied at all to 10=very satisfied
Patient global satisfaction | Day 56
  scale ranging from 0=not satisfied at all to 10=very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Marta Sar Pormian, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No